CLINICAL TRIAL: NCT01939587
Title: A Single-centre, Randomised, Double-blind, Placebo-controlled, 3-way Multiple Dose, Cross-over, "Proof-of-concept" Study to Assess the Efficacy of a Single PBF-680 Oral Administration to Attenuate Adenosine 5'-Monophosphate (AMP) Challenge-induced Airway Hyperresponsiveness in Mild-to-moderate Asthmatics
Brief Title: Study to Assess the Efficacy of a Single PBF-680 Oral Administration to Attenuate Adenosine 5'-Monophosphate Challenge-induced Airway Hyperresponsiveness in Mild-to-moderate Asthmatics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Palo Biofarma, S.L (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IIBSP-PBF-2013-93; 2013-002906-30 (EudraCT Number)
Record Dates: First submitted 2013-08-08; First posted 2013-09-11 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Asthma
Keywords: Adenosine A1 receptor antagonist; Asthma; adenosine receptor modulator; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PBF-680 5 mg (Experimental): 5 mg of PBF-680
  Interventions: Drug: PBF-680 5 mg
- PBF-680 20 mg (Experimental): 20 mg of PBF-680
  Interventions: Drug: PBF-680 20 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PBF-680 5 mg
  Arms: PBF-680 5 mg
Drug: PBF-680 20 mg
  Arms: PBF-680 20 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a single-center, double-blind, randomized trial utilizing a three-period, balanced block design, with each period comprising a unique study product administration. The treatments studied are PBF-680 5 mg, PBF-680 20 mg and placebo, as an orally administered capsule. The study includes a screening visit, a selection visit, three visits for the randomized treatment sequence, and an end-of-study follow-up visit, spanning through a 65-day maximum study duration. The study will be conducted on 18 male or female adults aged ³18 years, with a diagnosis of stable, mild to moderate asthma as per GINA guidelines, with no smoking or less than a 5 packs-years smoking history history, responsive to AMP airway challenge as determined in the selection visit.

The primary efficacy variable will be the PC20 yielded from AMP airway challenge testing at the three treatment visits. FeNO, sampled at three time points at each treatment period visit, will be a exploratory variable. Safety assessment will include monitoring of adverse events, physical examination, vital signs, EKGs, spirometry, serum and urine pregnancy tests, and laboratory determinations. Blood sampling at a time-point series will provide pharmacokinetics data.

The primary variable of the study is PC20, mg×mL-1. The PC 20 distributions will be analyzed by treatment using ANOVA for repeated measurements, followed by post hoc pairwise comparisons as appropriate. Other analyses will comprise FeNO, pharmacokinetics, data sets generated from baseline characteristics and safety assessments, and discretionary expiratory analyses to evaluate the influence of baseline and clinical covariates on the primary variable.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged 18, who have signed the informed consent form prior to initiation of any study procedures.
* Subjects with mild to moderate asthma, diagnosed as per Global Initiative for Asthma(GINA) guidelines.
* Subjects must have a body mass index between 18 and 35 kg/m².
* Subjects must be able to perform acceptable spirometry in accordance with ATS/ERS criteria for acceptability repeatability.
* Subjects must have a baseline FEV1 60% of predicted normal, and greater than 1 L in absolute value, on Visit 2.
* On Visit 2, eligible subjects must show airway hyperresponsiveness to AMP, determined by PC20 thresholding (the AMP provocative concentration that elicits a 20% drop from baseline FEV1 value, under AMP challenge test as per the ERS Task Force on Indirect Airway Challenges).

Exclusion Criteria:

* Current smokers, smokers within six months prior to Visit 1, or subjects with an smoking history greater than 5 pack-years.
* Asthmatics in treatment Step 5 as per GINA guidelines, including oral corticosteroids and/or omalizumab, or any immunosuppressive medication whether asthma-related or indicated for any concomitant morbidities.
* Subjects with a history of life-threatening asthma attacks (i.e. requiring ICU admission, orotracheal intubation).
* Subjects with a history of a respiratory tract infection or an asthma crisis requiring the use of antibiotics and/or systemic corticosteroids within 4 weeks prior to Visit 1, or who develop a respiratory tract infection or asthma crisis during the screening period. In the latter case, the subjects can be re-screened four weeks after the last dose of systemic corticosteroid or antibiotic.
* Subjects that received bronchial thermoplastic treatment.
* Subjects with concomitant pulmonary or thoracic disease other than asthma that could interfere safety or efficacy as per site investigator assessment. This includes, but is not limited to, COPD attributable to tobacco or alpha-1 antitrypsin deficiency, cystic fibrosis, sarcoidosis, interstitial lung disease, pulmonary hypertension, active pulmonary tuberculosis, or any prior condition that led to pulmonary resection surgery or lung transplantation. Non-cystic fibrosis bronchiectasis without clinically significant morbidity, moderate alpha-1 antitrypsin deficiency without evidence of emphysema or related COPD, or past pulmonary tuberculosis that received proper medical treatment, are acceptable provided that the condition is not expected to interfere with pulmonary function testing as per site investigator assessment.
* Subjects with symptoms of angina pectoris or with a history of confirmed coronary disease or cardiomyopathy.
* Subjects with A-V block in any degree, sinus bradycardia, tachyarrhythmia, unstable atrial fibrillation, long QT syndrome, QTc(F) interval greater than 450 ms at screening(Visit 2), or any other EKG abnormality deemed clinically significant by the investigator.
* Subjects who have a clinically significant laboratory abnormality at screening (Visit 2).
* Subjects with current uncontrolled arterial hypertension.
* Women of child-bearing potential, unless they are surgically sterile (i.e. bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy), are at least 2 years postmenopausal, practice abstinence, or agree to employ effective contraception from Visit 1 through Visit 6. Acceptable contraception procedures are oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, or use of a condom with spermicide by the sexual partner.
* Women supplying lactation.
* Receipt of any investigational drug therapy or biologicals within 3 months before randomization in this study, or within 5 half-lives of the investigational agent or biologic, whichever is longer.
* History of any known immunodeficiency disorder.
* Subjects with a history of malignancy within the past five years, with the exception of localized basal cell carcinoma of the skin.
* History of treatment for alcohol or drug abuse within the past year.
* Subjects with any comorbidity that could affect the safety or efficacy as per site investigator assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in PC20 yielded from AMP airway challenge testing | 2.25, 3.5, 8 hours post dose

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Palobiofarma S.L. (molecule owner), Mataró, Barcelona

REFERENCES:
- See also: Institut d'Investigació Biomèdica Sant Pau — http://www.iibsantpau.cat/
- See also: molecule owner — http://www.palobiofarma.com/